CLINICAL TRIAL: NCT02947750
Title: Neurovascular Regulation During Exercise in Humans With Chronic Kidney Disease
Brief Title: Neurovascular Transduction During Exercise in Chronic Kidney Disease
Acronym: NeurovEx
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeanie Park, Associate Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00091660; R01HL135183 (NIH)
Record Dates: First submitted 2016-10-17; First posted 2016-10-28 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Hypertension; Kidney Disorder; Nephrology; Physiology
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Kidney Diseases | interventions — sapropterin; Folic Acid; Exercise; Histidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Exercise training + 6R-BH4 (Experimental): Participants randomized to this arm will exercise on a stationary bicycle for 20-45 minutes, 3 times per week, for 6-12 weeks. This arm will also take the study drug 6R-BH4.
  Interventions: Drug: 6R-BH4; Dietary Supplement: Folic acid; Other: Exercise training
- Exercise training + 6R-BH4 placebo (Active Comparator): Participants randomized to this arm will exercise on a stationary bicycle for 20-45 minutes, 3 times per week, for 6-12 weeks. This arm will also take a placebo to match the study drug 6R-BH4.
  Interventions: Other: 6R-BH4 placebo; Dietary Supplement: Folic acid; Other: Exercise training
- Stretching + 6R-BH4 (Active Comparator): Participants randomized to this arm will do muscle stretching and toning for 20-45 minutes, 3 times per week, for 6-12 weeks. This arm will also take the study drug 6R-BH4.
  Interventions: Drug: 6R-BH4; Dietary Supplement: Folic acid; Other: Stretching
- Stretching + placebo (Placebo Comparator): Participants randomized to this arm will do muscle stretching and toning for 20-45 minutes, 3 times per week, for 6-12 weeks. This arm will also take a placebo instead of the active study drug.
  Interventions: Other: 6R-BH4 placebo; Dietary Supplement: Folic acid; Other: Stretching
- Exercise training + histidine and beta-alanine (Active Comparator): Participants randomized to this arm will exercise on a stationary bicycle for 20-45 minutes, 3 times per week, for 6-12 weeks. This arm will also take histidine and beta-alanine supplementation.
  Interventions: Other: Exercise training; Dietary Supplement: Histidine and beta-alanine supplementation
- Exercise training + histidine and beta-alanine placebo (Active Comparator): Participants randomized to this arm will exercise on a stationary bicycle for 20-45 minutes, 3 times per week, for 6-12 weeks. This arm will also take a placebo to match the histidine and beta-alanine supplementation.
  Interventions: Other: Exercise training; Other: Histidine and beta-alanine placebo

INTERVENTIONS:
Drug: 6R-BH4 — Participants will receive 200 mg of 6R-BH4 twice daily for 12 weeks. Study pills are dissolved in water or apple juice, and taken with food.
  Other Names: Tetrahydrobiopterin; Kuvan; Sapropterin dihydrochloride
  Arms: Exercise training + 6R-BH4; Stretching + 6R-BH4
Other: 6R-BH4 placebo — Participants will receive a placebo that is identical to 200 mg of 6R-BH4. The placebo will be taken twice daily for 12 weeks. Study pills are dissolved in water or apple juice, and taken with food.
  Arms: Exercise training + 6R-BH4 placebo; Stretching + placebo
Dietary Supplement: Folic acid — Participants will take 1 mg of folic acid daily for 12 weeks. Folic acid is given because it enhances the binding affinity of BH4 to nitric oxide synthase (NOS), and also enhances the regeneration of BH4 from inactive BH2
  Arms: Exercise training + 6R-BH4; Exercise training + 6R-BH4 placebo; Stretching + 6R-BH4; Stretching + placebo
Other: Exercise training — Participants will exercise 3 times a week on a stationary ergometer. Exercise intensity will begin at low levels (50% of maximal heart rate reserve) calculated utilizing the Karvonen method. Briefly, target exercise heart rate (HR) is calculated by subtracting the persons age from 220. Resting heart rate is then subtracted from this number. The answer is then multiplied by the target percent (50% for example) and the product is added back to resting heart rate to provide the target exercise session heart rate. Intensity will be increased by 5% every week (as tolerated by the participant) to a maximum of 80% of maximal heart rate. Exercise time will progress from an initial 20 minutes per session to a maximum of 45 minutes by increasing 5 minutes each week.
  Arms: Exercise training + 6R-BH4; Exercise training + 6R-BH4 placebo; Exercise training + histidine and beta-alanine; Exercise training + histidine and beta-alanine placebo
Other: Stretching — Participants randomized to 'No Exercise Training' group will instead of aerobic exercise, undergo progressive whole body stretching and toning exercises designed for individuals 65 and older. This type of low intensity activity is designed not to increase heart rate and will serve as the Control group to the Exercise Training group. The Control group will come in for stretching sessions 3 times per week for 20-45 minutes.
  Other Names: Control for exercise training
  Arms: Stretching + 6R-BH4; Stretching + placebo
Dietary Supplement: Histidine and beta-alanine supplementation — Histidine and beta-alanine are two over-the-counter supplements commonly used to enhance sports performance in athletes. Participants randomized to this study arm will receive combined histidine (4g/day) and beta-alanine (3.2g/day) supplementation.
  Arms: Exercise training + histidine and beta-alanine
Other: Histidine and beta-alanine placebo — Participants randomized to this study arm will receive a placebo to match combined histidine (4g/day) and beta-alanine (3.2g/day) supplementation.
  Arms: Exercise training + histidine and beta-alanine placebo

SUMMARY:
The purpose of this study is to find out why patients with chronic kidney disease (CKD) have poor exercise capacity and to explore what causes an increase in blood pressure during exercise (i.e. increased adrenaline levels, or decreased ability of blood vessels to dilate). This study will also test whether or not regular exercise on a bicycle and/or treatment with 6R-BH4 (Kuvan) pills, or histidine and beta-alanine supplementation improves these measures during exercise. 6R-BH4 is currently FDA-approved for use in patients with certain forms of a disease called phenylketonuria, but it is not currently FDA approved for blood pressure or exercise capacity in people with CKD.

DETAILED DESCRIPTION:
The major problem addressed in this study is to understand mechanisms underlying poor exercise capacity in patients with chronic kidney disease (CKD). Prior research has found that CKD patients have an exaggerated increase in blood pressure during certain forms of exercise that could contribute to exercise dysfunction as well as cardiovascular disease. This study will test the mechanisms underlying this exaggerated blood pressure response, as well as the potential benefits of simple measures such as exercise training on a stationary bicycle, and treatment with 6R-BH4, a drug that is currently FDA-approved for the treatment of phenylketonuria, but has been shown to have beneficial effects on vascular health in patients with kidney disease. This study will also examine the effects of exercise with histidine and beta-alanine supplementation. Histidine and beta-alanine are two over-the-counter supplements commonly used to enhance sports performance in athletes.

Prior to the intervention portion of this study, the researchers will measure how much the vein constricts in response to adrenaline in CKD patients versus controls. The study will also measure muscle pH, and muscle oxygenation during exercise in CKD patients and controls.

The intervention portion of the study will test whether aerobic exercise training with and without 6R-BH4, or with and without histidine and beta-alanine supplementation might help muscle pH and adrenaline levels, vascular reactivity, muscle oxygenation, and the exaggerated blood pressure response during exercise in CKD patients. Participants will be randomized using a 2x2 factorial design to exercise training (ET) with 6R-BH4, ET with placebo, stretching (control condition to exercise) with 6R-BH4, and stretching with placebo. Participants will undergo exercise training on a stationary bicycle, or stretching exercises, 3 times per week for 6-14 weeks (depending on availability of the participant).

ELIGIBILITY:
Inclusion Criteria for Chronic Kidney Disease Patients:

* Stage III or IV Chronic Kidney Disease, defined as reduction in estimated glomerular filtration rate (eGFR) to 15-59 cc/minute as calculated by the modified Modification of Diet in Renal Disease (MDRD) Study equation or the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* Stable renal function, with no greater than a 30% reduction in eGFR over the prior 3 months
* Does not exercise regularly (defined as exercising less than 20 minutes twice per week)
* Willing and able to cooperate with the study protocol

Inclusion Criteria for Control Study Participants:

* Does not exercise regularly (defined as exercising less than 20 minutes twice per week)
* Willing and able to cooperate with the study protocol

Exclusion Criteria:

* severe CKD (eGFR<15 cc/minute)
* ongoing drug or alcohol abuse
* diabetic neuropathy
* any serious systemic disease that might influence survival
* severe anemia with hgb level <9 g/dL
* clinical evidence of congestive heart failure or ejection fraction below 35%
* symptomatic heart disease determined by prior electrocardiogram, stress test, and/or history
* treatment with central alpha agonists (clonidine)
* uncontrolled hypertension with BP greater than 170/100 mm Hg
* low blood pressure with BP less than 100/50
* pregnancy or plans to become pregnant
* current treatment with monoamine oxidase (MAO) inhibitors
* inability to exercise on a stationary bicycle

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in functional sympatholysis | Baseline, Week 12
  Muscle oxygenation during exercise and sympathoexcitation will be measured.
Change in vascular alpha 1 adrenergic responsiveness | Baseline, Week 12
  Changes in vascular diameter in response to phenylephrine will be measured.
Change in exaggerated pressor responses during exercise | Baseline, Week 12
  Blood pressure and sympathetic responses during exercise will be measured.

SECONDARY OUTCOMES:
Renal artery resistance during exercise | Baseline, Week 12
  Renal artery blood flow will be measured.
Change in endothelial function | Baseline, Week 12
  Endothelial function using peripheral arterial tonometry will be measured.
Change in vascular stiffness | Baseline, Week 12
  Vascular stiffness using applanation tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Nocera, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta VA Health Care System, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeong J, Sprick JD, DaCosta DR, Mammino K, Nocera JR, Park J. Exercise modulates sympathetic and vascular function in chronic kidney disease. JCI Insight. 2023 Feb 22;8(4):e164221. doi: 10.1172/jci.insight.164221. PMID 36810250